CLINICAL TRIAL: NCT03453944
Title: Breath Synchronized Electrical Stimulation of the Abdominal Wall Muscles to Prevent Respiratory Muscle Atrophy During the Acute Stages of Mechanical Ventilation Therapy
Brief Title: NMES to Prevent Respiratory Muscle Atrophy in Mechanically Ventilated Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Medical Center Nijmegen (Other)
Collaborators: Liberate Medical (Industry); Amsterdam UMC, location VUmc (Other); Canisius-Wilhelmina Hospital (Other)
Responsible Party: Principal Investigator, Leo Heunks, MD, Prof, Amsterdam UMC, location VUmc
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: LM-RB-01
Record Dates: First submitted 2017-04-25; First posted 2018-03-05 (Actual); Last update posted 2018-03-05 (Actual); Status verified 2018-02

CONDITIONS: Mechanical Ventilation Complication; Neuromuscular Electrical Stimulation; Muscle Weakness
Keywords: Expiratory muscles; Mechanically ventilated patients; Neuromuscular electrical stimulation; Respiratory function; Ventilator-acquired muscle atrophy
MeSH Terms: conditions — Muscle Weakness; Respiratory Aspiration

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VF03-K active stimulation (Experimental): NMES applied to the abdominal wall muscles using the VentFree prototype (VF03-K). Stimulation is applied twice daily for 30 minutes, 5 days per week, for 6 weeks or until the patient is weaned from mechanical ventilation, whichever occurs sooner.
  Interventions: Device: VentFree prototype (VF03-K) active stimulation
- VF03-K sham stimulation (Sham Comparator): Sham stimulation applied to the abdominal wall muscles using the VentFree prototype (VF03-K). Sham stimulation is applied twice daily for 30 minutes, 5 days per week, for 6 weeks or until the patient is weaned from mechanical ventilation, whichever occurs sooner.
  Interventions: Device: VentFree prototype (VF03-K) sham stimulation

INTERVENTIONS:
Device: VentFree prototype (VF03-K) active stimulation — Abdominal wall muscle stimulation synchronised with mechanical ventilation. Stimulation frequency: 30 Hz, pulse width: 352us, max. intensity: 100mA (threshold intensity determined using ultrasound)
  Arms: VF03-K active stimulation
Device: VentFree prototype (VF03-K) sham stimulation — Abdominal wall muscle sham-stimulation synchronised with mechanical ventilation. Stimulation frequency: 10 Hz, pulse width: 352us, intensity: 15 mA.
  Arms: VF03-K sham stimulation

SUMMARY:
Patients requiring prolonged time on the ventilator are susceptible to a wide range of clinical complications and excess mortality. It is therefore imperative for them to wean at the earliest possible time.

Respiratory muscle weakness due to disuse of these muscles is a major underlying factor for weaning failure. Surprisingly, there is not much known about the impact of critical illness and MV on the expiratory abdominal wall muscles.These muscles are immediately activated as ventilation demands increase and are important in supporting respiratory function in patients with diaphragm weakness. Weakness of expiratory abdominal wall muscles will result in a decreased cough function and reduced ventilatory capacity. These are considerable causes of weaning failure and (re)hospitalisation for respiratory complications such as pneumonia.

Recent evidence shows that neuromuscular electrical stimulation (NMES) can be used as a safe therapy to maintain skeletal muscle function in critically ill patients. This study will be the first to test the hypothesis that breath-synchronized NMES of the abdominal wall muscles can prevent expiratory muscle atrophy during the acute stages of MV.

DETAILED DESCRIPTION:
Approximately 30-40% of intubated patients at the intensive care unit (ICU) take more than one attempt to wean from mechanical ventilation (MV). 6-14% of intubated patients take longer than 7 days to wean from MV. Patients requiring prolonged time on the ventilator are susceptible to a wide range of clinical complications and excess mortality. It is therefore imperative for them to wean at the earliest possible time.

Respiratory muscle weakness due to disuse of these muscles is a major underlying factor for weaning failure. It is known that diaphragm strength rapidly declines within a few days after the initiation of MV. Surprisingly, there is not much known about the impact of critical illness and MV on the expiratory abdominal wall muscles.These muscles are immediately activated as ventilation demands increase and are important in supporting respiratory function in patients with diaphragm weakness. Weakness of expiratory abdominal wall muscles will result in a decreased cough function and reduced ventilatory capacity. These are considerable causes of weaning failure and (re)hospitalisation for respiratory complications such as pneumonia.

Recent evidence shows that neuromuscular electrical stimulation (NMES) can be used as a safe therapy to maintain skeletal muscle function in critically ill patients, e.g. by stimulating quadriceps muscles in patients receiving MV.

This study will be the first to test the hypothesis that exhalation synchronized NMES of the abdominal wall muscles can prevent expiratory muscle atrophy during the acute stages of MV. The investigators hypothesize that this approach will improve respiratory function and thereby will reduce the amount of time it takes to wean patients from mechanical ventilation.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 year
* invasive mechanical ventilation less than 72 hours
* expected duration of MV after inclusion > 72 hours

Exclusion Criteria:

* no clearly visible separate layers of the abdominal wall muscles (external oblique, internal oblique and transverse abdominal muscles), assessed with ultrasound during routine care
* cardiac pacemaker
* congenital myopathies and/or existing central or peripheral neuropathies
* refractory epilepsy
* recent abdominal surgery within four weeks prior to study inclusion
* body mass index (BMI) greater than 35 kg/m2
* pregnancy

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-03-09 (Actual); Primary Completion 2018-07-01 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
Thickness of the abdominal wall muscles | Until study completion, up to 6 weeks
  Thickness of the abdominal wall muscles over time, for both groups, as measured by ultrasound.

SECONDARY OUTCOMES:
Thickness of the diaphragm | Until study completion, up to 6 weeks
  Thickness of the diaphragm over time, for both groups, as measured by ultrasound.
Thickness of the rectus abdominis muscle | Until study completion, up to 6 weeks
  Thickness of the rectus abdominis mucle over time, for both groups, as measured by ultrasound.
Maximum expiratory pressure (MEP) | Within 24 hours after extubation
  Maximum expiratory pressure (MEP) to assess expiratory muscle function
Maximum inspiratory pressure (MIP) | Within 24 hours after extubation
  Maximum inspiratory pressure (MIP) to assess inspiratory muscle function
Vital capacity (Vc) | Within 24 hours after extubation
  Vital capacity (Vc) to assess respiratory muscle strength
Peak expiratory flow | Within 24 hours after extubation
  Peak expiratory flow (PEF) to assess cough strength
Number of patients with extubation failure | Within 24 hours after extubation
  Weaning failure defined as the failure to pass a spontaneous-breathing trial or the need for reintubation within 48 hours following extubation
Systemic inflammatory markers | Within 24 hours after extubation
  Among others, cytokines IL-6 and IL-1 will be determined from blood sample analysis
Number of patients with respiratory complications after ICU discharge | Up to 6 weeks after ICU discharge
  Number of patients with development of pneumonia, and readmission to the ICU due to atelectasis or respiratory problems that require mechanical ventilation.

OTHER OUTCOMES:
Expiratory flow limitation (optional) | Measured before the first NMES session and within 24 hours after extubation
  EFL test to determine flow limitation in COPD

CONTACTS AND LOCATIONS:
Overall Officials: Angelique ME Spoelstra-de Man, MD, PhD, Principal Investigator — Amsterdam UMC, location VUmc
Locations (3):
- Netherlands (3):
  - UMC Nijmegen, Nijmegen, Gelderland
  - Canisius Wilhelmina Hospital, Nijmegen, Gelderland
  - VU University Medical Center, Amsterdam, North Holland

REFERENCES:
- [Derived] Jonkman AH, Frenzel T, McCaughey EJ, McLachlan AJ, Boswell-Ruys CL, Collins DW, Gandevia SC, Girbes ARJ, Hoiting O, Kox M, Oppersma E, Peters M, Pickkers P, Roesthuis LH, Schouten J, Shi ZH, Veltink PH, de Vries HJ, Shannon Weickert C, Wiedenbach C, Zhang Y, Tuinman PR, de Man AME, Butler JE, Heunks LMA. Breath-synchronized electrical stimulation of the expiratory muscles in mechanically ventilated patients: a randomized controlled feasibility study and pooled analysis. Crit Care. 2020 Oct 30;24(1):628. doi: 10.1186/s13054-020-03352-0. PMID 33126902